CLINICAL TRIAL: NCT04252820
Title: Prevention of Perioperative Hypothermia in Transurethral Resection Under Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra, Principal Investigator, Anesthesiologist, Dr. Negrin University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RTU-Spinal
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Hypothermia; Anesthesia; Perioperative Complication; Regional Anesthesia Morbidity; Temperature Change, Body; Transurethral Resection Syndrome
Keywords: body temperature; hypothermia; prewarming; regional anesthesia
MeSH Terms: conditions — Hypothermia; Body Temperature Changes; Transurethral resection syndrome

STUDY DESIGN:
Intervention Model Description: Different time periods of prewarming will be compared: 0 minutes (control group), 15 minutes, 30 minutes and 45 minutes
Who Masked: Care Provider, Investigator
Masking Description: Randomization will be carried out by a collaborator investigator using a computer program (Excel 2016) when a new patient is included into the clinical trial. This collaborator investigator will tell the nurse in charge of receiving the patient in the preanesthetic room how long prewarming has to be given to the patient: 0 minutes (no prewarming), 15 minutes, 30 minutes or 45 minutes, according to the group given by the computer program. This collaborator investigator will not provide clinical care to the patient. Attending anesthesiologist will be blind to the allocation of the participants. Principal investigator will not be able to know how long prewarming will be given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No prewarming. Patients will be actively warmed during the intraoperative period. Tympanic thermometer and zero-heat-flux temperature sensor will be used to measure the temperature throughout the perioperative period.
- Prewarming during 15 minutes (Experimental): Active Prewarming will be performed during 15 minutes, using a forced-air blanket over the whole body and connected to a forced-air warmer set up at 43 degrees centigrade. Patients will be actively warmed during the intraoperative period.
  Interventions: Device: WarmTouch total body blanket, Covidien Ltd, Mansfield, USA
- Prewarming during 30 minutes (Experimental): Active Prewarming will be performed during 30 minutes, using a forced-air blanket over the whole body and connected to a forced-air warmer set up at 43 degrees centigrade. Patients will be actively warmed during the intraoperative period.
  Interventions: Device: WarmTouch total body blanket, Covidien Ltd, Mansfield, USA
- Prewarming during 45 minutes (Experimental): Active Prewarming will be performed during 45 minutes, using a forced-air blanket over the whole body and connected to a forced-air warmer set up at 43 degrees centigrade. Patients will be actively warmed during the intraoperative period.
  Interventions: Device: WarmTouch total body blanket, Covidien Ltd, Mansfield, USA

INTERVENTIONS:
Device: WarmTouch total body blanket, Covidien Ltd, Mansfield, USA — Forced-air warming will be applied in the preanesthetic room
  Arms: Prewarming during 15 minutes; Prewarming during 30 minutes; Prewarming during 45 minutes

SUMMARY:
Perioperative hypothermia is one of the most common anaesthetic complications, increasing the morbidity/mortality of our patients. Active prewarming with hot forced-air devices has demonstrated to be the most effective tool to prevent hypothermia, but its use is only recommended in long-term surgeries and the optimal prewarming duration has not been elucidated. Both spinal anaesthesia associated to the irrigation with liquids at low temperature instilled during transurethral resection (TUR) cause a decrease in the core temperature of the patient. This is a clinical trial comparing different time periods of prewarming in patients submitted to undergo elective transurethral resection. Our aim is to assess the effect of different time-periods of prewarming on preventing perioperative hypothermia during TUR with spinal anaesthesia. Investigators will compare different time periods: 0 minutes (control group), 15 minutes, 30 minutes and 45 minutes. 200 patients are going to be included in this study (50 patients in each group). Measurement of temperature will be performed using a tympanic thermometer and zero-heat-flux temperature sensor. Patients will be followed throughout their hospital admission. Data will be recorded using a validated instrument and will be analysed using the statistics program R Core Team.

DETAILED DESCRIPTION:
Inadvertent perioperative hypothermia is probably the most common anaesthetic complication. Its appearance increases the morbidity of the surgical patient, increasing the incidence of cardiac events or perioperative blood loss and causes a greater time of recovery from anaesthesia. Prewarming is the most effective measure to prevent hypothermia and maintain intraoperative normothermia. However, prewarming in patients submitted to spinal anesthesia is still a weak recommendation and the optimal prewarming time has not been elucidated. Due to the searching of optimal prewarming time and the lack of evidence about the efficiency of prewarming in patients submitted to transurethral resection under spinal anaesthesia, the conductance of this clinical trial is justified.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective Transurethral resection under spinal anesthesia.
* Patients older tan 18 years old.
* American Society of Anesthesiologists physical status classification I - III.
* Absence of cognitive impairment.
* Written informed consent before enrollment.

Exclusion Criteria:

* Pregnancy.
* American Society of Anesthesiologists physical status classification IV.
* Active infection.
* Intake of antipyretics within 24 hours before surgery.
* Thyroid disorders.
* Skin lesions or History of hypersensitivity to skin contact devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Differences in Body Temperature among different treatment groups using tympanic thermometer and zero-heat-flux temperature sensor | Throughout surgery, an average of 60 minutes.
  To assess the effects of prewarming in preventing drop of body temperature of patients undergoing elective transurethral resection under spinal anesthesia

SECONDARY OUTCOMES:
Length of stay in postanesthetic care unit (in minutes) | Stay in Post-Anesthetic Care Unit, an average of 6 hours.
  To assess the effect of prewarming in the length of stay in the Post-Anesthetic Care Unit of patients undergoing elective transurethral resection under spinal anesthesia.
Postoperative pain, using visual analogue scale (from 0 to 10) | Immediate postoperative period, an average of 1 hour.
  To assess the effect of prewarming in reducing the postoperative pain at the arrival to the postanesthetic care unit of patients undergoing elective transurethral resection under spinal anesthesia
Postoperative shivering (using a dichotomous scale: yes or no) | Immediate postoperative period, an average of 1 hour
  To assess the effect of prewarming in the prevalence of postoperative shivering of patients undergoing elective transurethral resection under spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Rodríguez-Pérez, PhD, Study Director — Dr Negrin UH
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data are to be shared with other researchers when required once the study is completed and global data are published.